CLINICAL TRIAL: NCT01022281
Title: Evaluation of Scanning Laser Polarimetry Findings in Individuals With Exfoliation Syndrome Compared With Normal Controls
Brief Title: Early Diagnosis in Glaucoma With GDxVcc
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Other Study IDs: A3631
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Exfoliation Syndrome
Keywords: Exfoliation; Scanning Laser Polarimetry; Corneal Thickness
MeSH Terms: conditions — Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Controls: Normal age matched controls without exfoliation
- Exfoliation Syndrome: Patients with exfoliation syndrome

SUMMARY:
To compare the Retina Nerve Fiber Layer thickness, measured with Scanning Laser Polarimetry in subjects with exfoliation syndrome and normal controls and to evaluate the value of scanning laser polarimetry in the early diagnosis and management of exfoliative glaucoma

DETAILED DESCRIPTION:
To compare the Scanning Laser Polarimetry findings in subjects with exfoliation syndrome and normal controls and to evaluate the value of scanning laser polarimetry in the early diagnosis and management of exfoliative glaucoma. Prospective study in progress. The investigators compare and analyze the scanning laser polarimetry parameters in consecutive subjects with exfoliation syndrome and normal intraocular pressure and compared them with consecutive normal controls. Randomly selected patients with exfoliation syndrome and normal controls undergo a comprehensive ophthalmic exam which includes 3 IOP measurements, corneal pachymetry, automated perimetry and assessment of the retina nerve fiber layer with scanning laser polarimetry. The investigators hypothesize that patients with exfoliation syndrome may show worse scanning laser polarimetry parameters than normal controls and this may prove to be an early sign of exfoliative glaucoma development. Evaluation of retina nerve fiber layer thickness may help us in identifying earlier those individuals with exfoliation syndrome that will develop exfoliative glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Exfoliation material on pupil
* Intraocular pressure below 21 mm Hg without therapy
* No glaucomatous damage
* Age between 60-75
* Open angle

Exclusion Criteria:

* Other Ophthalmic diseases
* Dry eye
* Corneal disorders
* Diabetic Retinopathy
* Optic Neuropathy (other than glaucomatous neuropathy)
* Ocular surgery or laser

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with and without exfoliation
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Scanning laser polarimetry parameters, evaluation of retina nerve fiber layer thickness | Morning measurement (10:00 - 13:00)

SECONDARY OUTCOMES:
Corneal thickness, exfoliation syndrome subjects that will develop exfoliation glaucoma | 10:00-13:00

CONTACTS AND LOCATIONS:
Overall Officials: Antonios T Dimopoulos, MD, Study Director — 1st University Department of Ophthalmogy
Locations (1):
- Glaucoma Unit, 1st University Department of Ophthalmology, Thessaloniki, Greece